CLINICAL TRIAL: NCT03560583
Title: Efficacy of Metoclopramide in Poor Ovarian Response IVF Patients: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Metoclopramide in Poor Ovarian Response IVF Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Leon Grin, Gynecological Doctor, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRZ 0046-17 CTIL
Record Dates: First submitted 2018-06-07; First posted 2018-06-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Poor Responders in IVF
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoclopramide 10 mg BID (Experimental)
  Interventions: Drug: Metoclopramide
- Placebo 10 mg BID (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metoclopramide — Metoclopramide 10 mg BID
  Arms: Metoclopramide 10 mg BID
Drug: Placebo Oral Tablet — Placebo 10 mg BID
  Arms: Placebo 10 mg BID

SUMMARY:
Poor ovarian response population of ART are considered the biggest challenge for providers. Hitherto, no one protocol has been proven to be effect in this subgroup of IVF patients.

Metoclopramide belongs to the antiemetic group, used for motion sickness and during early gestation for hyperemesis gravidarum.

The mechanism of action is antagonisim to dopamine receptors. We hypothesize than by blocking dopamine receptors and decreasing the dopaminergic tone there is a possibility to increase the sensitivity of ovarian response to gonadotropins during controlled ovarian stimulation and result in increased oocyte retrival.

ELIGIBILITY:
Inclusion Criteria:

* Poor response according to "Bologna criteria"

Exclusion Criteria:

* Allergy to metoclopramide
* Prolactinemia
* Women treated with dopamine agonists

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 60 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes | Approximately 5 weeks from first dose of study drug
  Number of oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Leon Grin, MD, Principal Investigator — Barzilai Medical Center
Locations (1):
- Barzilai University Medical Center, Ashkelon, Ashkelon District, Israel

REFERENCES:
- [Background] Boelig RC, Barton SJ, Saccone G, Kelly AJ, Edwards SJ, Berghella V. Interventions for treating hyperemesis gravidarum: a Cochrane systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2018 Sep;31(18):2492-2505. doi: 10.1080/14767058.2017.1342805. Epub 2017 Jul 11. PMID 28614956
- [Background] Hernandez I, Parra A, Mendez I, Cabrera V, Cravioto MC, Mercado M, Diaz-Sanchez V, Larrea F. Hypothalamic dopaminergic tone and prolactin bioactivity in women with polycystic ovary syndrome. Arch Med Res. 2000 Mar-Apr;31(2):216-22. doi: 10.1016/s0188-4409(00)00059-x. PMID 10880731
- [Background] Prelevic GM, Wurzburger MI, Peric LA. Metoclopramide effect on serum prolactin LH and FSH in patients with polycystic ovary syndrome. J Endocrinol Invest. 1988 Apr;11(4):255-9. doi: 10.1007/BF03350148. PMID 3137253
- [Background] Mendes MC, Ferriani RA, Sala MM, Moura MD, Carrara HH, de Sa MF. Effect of transitory hyperprolactinemia on in vitro fertilization of human oocytes. J Reprod Med. 2001 May;46(5):444-50. PMID 11396370